CLINICAL TRIAL: NCT05094336
Title: A Phase 1/1b/2 Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of AMG 193 Alone and in Combination With Docetaxel in Subjects With Advanced MTAP-null Solid Tumors
Brief Title: A Study of AMG 193 in Participants With Advanced MTAP-null Solid Tumors (MTAPESTRY 101)
Acronym: MTAPESTRY 101
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20210023; 2023-504363-17 (Other: EU CT Number)
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced MTAP-null Solid Tumors
Keywords: Metastatic MTAP-null solid tumors; Advanced MTAP-null solid tumors; Non-small cell lung cancer; Biliary Tract Cancer (BTC); Head and neck squamous cell carcinoma; Pancreatic adenocarcinoma; Esophageal cancer; Gastric cancer; Glioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Biliary Tract Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esophageal Neoplasms; Stomach Neoplasms; Glioma | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part 1a, Phase 1: AMG 193 Monotherapy Dose Exploration (Experimental): Participants with MTAP-null solid tumors will receive escalating doses of AMG 193 to estimate the MTD and/or the RP2D.
  Interventions: Drug: AMG 193
- Part 1c, Phase 1: AMG 193 Monotherapy Dose Expansion (Experimental): Participants will receive the identified MTD/RP2D of AMG 193 in the following cohort: MTAP-null NSCLC.
  Interventions: Drug: AMG 193
- Part 2a, Phase 1: AMG 193 Dose Exploration + Docetaxel (Experimental): Participants with MTAP-null NSCLC will receive escalating doses of AMG 193 + a fixed dose of docetaxel to estimate the MTD/RP2D of the combination.
  Interventions: Drug: AMG 193; Drug: Docetaxel
- Part 2b, Phase 1: AMG 193 + Docetaxel Dose Expansion (Experimental): Participants with MTAP-null NSCLC will receive the identified MTD/RP2D of AMG 193 + docetaxel.
  Interventions: Drug: AMG 193; Drug: Docetaxel
- Part 3: AMG 193 Phase 2 (Experimental): Participants with MTAP-null solid tumors will receive AMG 193.
  Interventions: Drug: AMG 193
- Part 1e, Phase 1: AMG 193 Monotherapy Dose Expansion (Experimental): Participants will receive the identified selected dose/MTD of AMG 193 in the following cohort: MTAP-null BTC.
  Interventions: Drug: AMG 193
- Part 1f, Phase 1: AMG 193 Monotherapy Dose Expansion (Experimental): Participants will receive the identified selected dose/MTD of AMG 193 in the following cohort:
  MTAP-null head and neck squamous cell carcinoma (HNSCC).
  Interventions: Drug: AMG 193
- Part 1g, Phase 1: AMG 193 Monotherapy Dose Expansion (Experimental): Participants will receive the identified selected dose/MTD of AMG 193 in the following cohort:
  MTAP-null pancreatic adenocarcinoma.
  Interventions: Drug: AMG 193
- Part 1h, Phase 1: AMG 193 Monotherapy Dose Expansion (Experimental): Participants will receive the identified selected dose/MTD of AMG 193 in the following cohort: MTAP-null or lost MTAP expression solid tumors (other than lymphoma or primary brain tumor).
  Interventions: Drug: AMG 193
- Part 1i, Phase 1: AMG 193 Dose Optimization (Experimental): Participants will receive a randomized dose optimization evaluation of AMG 193.
  Interventions: Drug: AMG 193
- Part 1j, Phase 1: AMG 193 DSPS Substudy (US Sites Only) (Experimental): Participants will receive doses of AMG 193 and comparator AMG 193 test tables at different times in a fasted state.
  Interventions: Drug: AMG 193; Drug: Comparator AMG 193 Test Tablet
- Part 1k, Phase 1: AMG 193 Food Effect Substudy (US Sites Only) (Experimental): Participants will receive AMG 193 once on a fasted state and once after eating a standardized high-fat, high calorie meal.
  Interventions: Drug: AMG 193
- Part 1l, Phase 1: AMG 193 Monotherapy Dose Expansion (Experimental): Participants will receive the identified selected dose/MTD of AMG 193 in the following cohort: MTAP-null esophageal/gastric cancer.
  Interventions: Drug: AMG 193
- Part 1m, Phase 1: AMG 193 Monotherapy Dose Expansion (Experimental): Participants will receive the identified selected dose/MTD of AMG 193 in the following cohort: MTAP-null glioma.
  Interventions: Drug: AMG 193

INTERVENTIONS:
Drug: AMG 193 — AMG 193: Orally via tablet
  Other Names: MTA Cooperative PRMT5 inhibitor
Drug: Docetaxel — Docetaxel: Intravenous infusion
  Arms: Part 2a, Phase 1: AMG 193 Dose Exploration + Docetaxel; Part 2b, Phase 1: AMG 193 + Docetaxel Dose Expansion
Drug: Comparator AMG 193 Test Tablet — Comparator AMG 193 test tablet: Orally via tablet. Only participants in the DSPS group of the Part 1a, Phase 1: AMG 193 Monotherapy Dose Exploration, and Part 1j, Phase 1 arms will receive comparator AMG 193 test tablet.
  Arms: Part 1j, Phase 1: AMG 193 DSPS Substudy (US Sites Only)

SUMMARY:
The primary objective of Parts 1 and 2 of this study is to evaluate the safety, tolerability, and to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of AMG 193 alone and in combination with docetaxel in adult participants with metastatic or locally advanced methylthioadenosine phosphorylase (MTAP)-null solid tumors.

The primary objective of Part 3 of this study is to evaluate the efficacy of AMG 193 in adult participants with metastatic or locally advanced MTAP-null solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent before initiation of any study specific activities/procedures.
* Age ≥ 18 years.
* Evidence of homozygous loss of cyclin dependent kinase inhibitor 2A (CDKN2A) (null) (Parts 1a, 1j, 1k, and 2a only) and/or methylthioadenosine phosphorylase (MTAP) (null) in the tumor tissue or blood (Parts 1a to 1k, Parts 2a and 2b) or lost MTAP expression in the tumor tissue (Parts 1a to 1k, Parts 2a and 2b).
* Histologically confirmed metastatic or locally advanced solid tumor not amenable to curative treatment with surgery and/or radiation.
* Able to swallow and retain orally (PO) administered study treatment and willing to record daily adherence to investigational product.
* Disease measurable as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Note: except participants enrolling to Part 1m.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Adequate hematopoietic function per local laboratory
* Adequate renal function per local laboratory
* Adequate glucose control per local laboratory (Part 1 only)
* Adequate liver function per local laboratory
* Adequate coagulation parameters
* Adequate pulmonary function
* Adequate cardiac function
* Minimum life expectancy of 12 weeks as per investigator judgement.
* Archived tumor tissue (formalin-fixed, paraffin-embedded [FFPE] sample collected within 5 years) or an archival block must be available.
* For Part 1f (MTAP-null or lost MTAP expression HNSCC): Must be willing to undergo tumor biopsy.
* For Part 1a: Must be willing to undergo tumor biopsy, before start of treatment (archival sample acceptable if obtained with 6 months of enrollment and subject has not received any other treatment since sample was obtained) and while on treatment.
* For DSPS study (Part 1j): Must be willing to participate in DSPS substudy (US sites only).

Food Effect Substudy (Part 1k): Specific Inclusion Criteria

* Subject able and willing to eat a standardized high-fat, high-caloric meal
* Subject able and willing to fast for ≥ 6 hours

Specific Inclusion Criteria for subjects with glioma (Part 1m only)

- Disease measurable as defined per Modified Response Assessment in Neuro-Oncology Criteria 2.0 (mRANO 2.0)

Exclusion Criteria:

* Spinal cord compression or untreated brain metastases or leptomeningeal disease.
* History of other malignancy within the past 2 years
* Any evidence of current interstitial lung disease
* Active infection
* Evidence of active severe acute respiratory syndrome coronavirus 2 (SARS-COV2) infection.
* History of arterial thrombosis
* Myocardial infarction and/or symptomatic congestive heart failure.
* Gastrointestinal tract disease
* History of bowel obstruction, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
* History of solid organ transplant.
* Diagnosis of Congenital Short QT Syndrome.
* Major surgery
* Anti-tumor therapy within 28 days of study day 1.
* Prior treatment with an methionine adenosyltransferase 2α (MAT2A) inhibitor or a protein arginine methyltransferase 5 (PRMT5) inhibitor.
* Prior treatment with docetaxel (Part 2 only)
* Prior irradiation to 25% of the bone marrow.
* Therapeutic or palliative radiation therapy within 2 weeks of study day 1.
* Live vaccine therapy within 4 weeks before study drug administration.
* Use of therapeutic anti-coagulation for treatment of active thromboembolic events.
* Use of prescription medications that are known strong inducers of cytochrome P450 3A4 (CYP3A4) within 14 days or 5 half-lives (whichever is longer) before study day 1
* Unresolved toxicity from prior anti-cancer therapy
* Currently receiving treatment in another investigational device or drug study.
* Known positive test for Human Immunodeficiency Virus (HIV).
* Positive hepatitis B surface antigen
* positive hepatitis C virus ribonucleic acid (RNA) by polymerase chain reaction (PCR)
* Female participants of childbearing potential unwilling to use protocol specified method of contraception

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2: Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) | 28 days
Parts 1 and 2: Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Up to approximately 3 years
  Adverse events (AEs) are defined as any untoward medical occurrence in clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurs after the participant has received study treatment. Any clinically significant changes in vital signs, electrocardiograms (ECGs) and clinical laboratory tests will be recorded as TEAEs.
  Serious AEs (SAEs) are defined as any event that meets at least 1 of the following serious criteria:
  * Results in death (fatal)
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other medically important serious event
Part 3: Objective Response Rate (ORR) | Up to approximately 3 years

SECONDARY OUTCOMES:
Parts 1 and 2: Maximal Plasma Concentration (Cmax) of AMG 193 | Cycle 1 Day 1 to Pre-Dose Cycle 5 Day 1 (Part 1 Cycle = 28 days, Part 2 Cycle =21 days)
Parts 1 and 2: Time to Achieve Maximal Plasma Concentration (Tmax) of AMG 193 | Cycle 1 Day 1 to Pre-Dose Cycle 5 Day 1 (Part 1 Cycle = 28 days, Part 2 Cycle =21 days)
Parts 1 and 2: Area Under the Plasma Concentration Versus Time Curve (AUC) of AMG 193 | Cycle 1 Day 1 to Pre-Dose Cycle 5 Day 1 (Part 1 Cycle = 28 days, Part 2 Cycle =21 days)
Part 2 Only: Maximal Plasma Concentration (Cmax) of Docetaxel | Cycle 1 Day 1 to Pre-Dose Cycle 5 Day 1 (Cycle =21 days)
Part 2 Only: Time to Achieve Maximal Plasma Concentration (Tmax) of Docetaxel | Cycle 1 Day 1 to Pre-Dose Cycle 5 Day 1 (Cycle =21 days)
Part 2 Only: Area Under the Plasma Concentration Versus Time Curve (AUC) of Docetaxel | Cycle 1 Day 1 to Pre-Dose Cycle 5 Day 1 (Cycle =21 days)
Parts 1 and 2: ORR | Up to approximately 3 years
Parts 1, 2 and 3: Disease Control Rate (DCR) | Up to approximately 3 years
Parts 1, 2 and 3: Duration of Response (DoR) | Up to approximately 3 years
Parts 1, 2 and 3: Time to Response (TTR) | Up to approximately 3 years
Parts 1, 2 and 3: Duration of Disease Control (DC) | Up to approximately 3 years
Parts 1, 2 and 3: Progression-Free Survival (PFS) | Up to approximately 3 years
Parts 1, 2 and 3: Overall Survival (OS) | Up to approximately 5 years
Part 3 Only: Number of Participants Who Experience TEAE | Up to approximately 3 years
  AEs are defined as any untoward medical occurrence in clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurs after the participant has received study treatment. Any clinically significant changes in vital signs, ECGs and clinical laboratory tests will be recorded as TEAEs.
  SAEs are defined as any event that meets at least 1 of the following serious criteria:
  * Results in death (fatal)
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other medically important serious event
Part 1a Only: Maximal Plasma Concentration (Cmax) of AMG 193 | Cycle 2 Day 1 to pre-dose on Cycle 2 Day 2 (Cycle = 28 days)
Part 1a Only: Time to Achieve Maximal Plasma Concentration (Tmax) of AMG 193 | Cycle 2 Day 1 to pre-dose on Cycle 2 Day 2 (Cycle = 28 days)
Part 1a Only: Area Under the Plasma Concentration Versus Time Curve (AUC) of AMG 193 | Cycle 2 Day 1 to pre-dose on Cycle 2 Day 2 (Cycle = 28 days)
Part 1a Only: Maximal Plasma Concentration (Cmax) of Comparator AMG 193 Test Tablet | Cycle 2 Day 2 to pre-dose on Cycle 2 Day 3 (Cycle = 28 days)
Part 1a Only: Time to Achieve Maximal Plasma Concentration (Tmax) of Comparator AMG 193 Test Tablet | Cycle 2 Day 2 to pre-dose on Cycle 2 Day 3 (Cycle = 28 days)
Part 1a Only: Area Under the Plasma Concentration Versus Time Curve (AUC) of Comparator AMG 193 Test Tablet | Cycle 2 Day 2 to pre-dose on Cycle 2 Day 3 (Cycle = 28 days)
Part 1k Only: Cmax of AMG 193 during fasted state | Cycle 2 day 1 pre-dose up to 24 hours post-dose (Cycle = 28 days)
Part 1k Only: Tmax of AMG 193 during fasted state | Cycle 2 day 1 pre-dose up to 24 hours post-dose (Cycle = 28 days)
Part 1k Only: AUC of AMG 193 during fasted state | Cycle 2 day 1 pre-dose up to 24 hours post-dose (Cycle = 28 days)
Part 1k Only: Cmax of AMG 193 during fed state | Cycle 2 day 2 pre-dose up to 24 hours post-dose (Cycle = 28 days)
Part 1k Only: Tmax of AMG 193 during fed state | Cycle 2 day 2 pre-dose up to 24 hours post-dose (Cycle = 28 days)
Part 1k Only: AUC of AMG 193 during fed state | Cycle 2 day 2 pre-dose up to 24 hours post-dose (Cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (75):
- United States (30):
  - City of Hope National Medical Center, Duarte, California
  - California Research Institute, Glendale, California
  - Fomat Medical Research, Oxnard, California
  - University of California at SF, San Francisco, California
  - D and H Cancer Research Center, Margate, Florida
  - Boca Raton Clinical Research Medical Center Inc, Tamarac, Florida
  - Goshen Health Systems, Goshen, Indiana
  - Indiana University, Indianapolis, Indiana
  - Community Health Network MD Anderson Cancer Center - North, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - American Oncology Partners, PA, Bethesda, Maryland
  - Henry Ford Cancer Detroit (Brigitte Harris Cancer Pavilion), Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health Monter Cancer Center, Lake Success, New York
  - New York University Grossman School of Medicine and New York University Langone Hospitals, New York, New York
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sanford Oncology Clinic and Pharmacy, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Dallas, Texas
  - Center for Oncology and Blood Disorders, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Lumi Research, Kingwood, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specialists PC, Fairfax, Virginia
- Australia (3):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Epworth Healthcare, East Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Parkville, Victoria
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (5):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (5):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
- France (4):
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Hopitaux Universitaires Pitie Salpetriere - Charles Foix, Paris
  - Gustave Roussy, Villejuif
- Germany (4):
  - Universitaetsklinikum Halle - Saale, Halle
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Japan (3):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Switzerland (5):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Universitaetsspital Zuerich, Zurich
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com